CLINICAL TRIAL: NCT00712413
Title: Pilot Study Assessing the Safety, Tolerability, Compliance and Efficacy of Twice Daily Dosed Pylera Plus Omeprazole as a First Line Treatment of Helicobacter Pylori Infection
Brief Title: Safety, Efficacy of Pylera BID Dosing in Eradication of H. Pylori
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PYLHp08-01
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori infection; Quadruple therapy; Safety; Efficacy; Tolerability; BID dosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: OBMT — Omeprazole 20 mg twice daily, in combination with bismuth subcitrate potassium (40 mg), metronidazole 125 mg and tetracycline 125 mg HCl. All patients must take 6 capsules of Pylera, in addition to 1 omeprazole twice daily
  Other Names: Pylera

SUMMARY:
The purpose of this study is to evaluate the effect of Pylera when given twice a day. Pylera approved treatment schedule is 3 pills taken 4 times daily, in addition to omeprazole given twice daily. In this trial, subjects with confirmed Helicobacter Pylori infection will receive Pylera treatment and omeprazole twice daily.

DETAILED DESCRIPTION:
This study will include three phases: screening, treatment and follow-up.

Screening: this phase will last a maximum of 15 days and subjects eligibility will be evaluated after informed consent signature. Urea breath test (UBT) will be performed in addition to routine baseline evaluations (physical, lab test, etc).

Treatment: subjects will be treated for 10 days. A "confirmation of eligibility" visit will take place on Day 0 and an "end-of-treatment" visit will take place between days 9-14.

Follow-up: approximately one month post-treatment, eradication of H. pylori will be confirmed through UBT

ELIGIBILITY:
Inclusion Criteria:

* Positive H. pylori status through UBT testing

Exclusion Criteria:

* Documented allergy to any of the drugs contained in the treatment regimen
* Severe renal insufficiency, renal failure or azotemia
* Previous surgery of the upper gastrointestinal tract
* Hepatic failure
* Pre-existing peripheral neuropathies
* Use of any experimental drug within 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
H. pylori status confirmed by Urea Breath Test | at 6 and 10 weeks following treatment

SECONDARY OUTCOMES:
Tolerability | at the end of treatment, one and two months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Monique Giguère, PhD, Study Director — Axcan Pharma inc
Locations (3):
- United States (2):
  - University of Michigan Health System, Ann Arbor, Michigan
  - Aurora Health Care, Milwaukee, Wisconsin
- McMaster University Medical Center, Division of Gastroenterology, Hamilton, Ontario, Canada